CLINICAL TRIAL: NCT06527040
Title: Clinical Decision Support for Safety of Opioid Transitions
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-1192; R61DA057610 (NIH)
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Medication Abuse; Harm Reduction
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Control group of contemporary encounters where clinical decision support alert is not active. Usual care.
- Clinical Decision Support (CDS): Opioid transition alert: Encounters where the opioid transition clinical decision support (CDS) alert fired. CDS logic is programmed to fire the alert when a provider places an order for an opioid that will transition the patient from acute to subacute opioid therapy (at 30 days) or from subacute to chronic opioid therapy (at 90 days).
  Interventions: Other: Opioid Transitions Clinical Decision Support (CDS)

INTERVENTIONS:
Other: Opioid Transitions Clinical Decision Support (CDS) — Clinical decision support in the form of an electronic health record (EHR) integrated, provider-facing alert suggesting (a) the patient is transitioning to a new phase of opioid therapy and (b) the provider should review patient pain data and pain management goals as suggested by Center for Disease Control and Prevention (CDC) guidelines.
  Groups: Clinical Decision Support (CDS): Opioid transition alert

SUMMARY:
The objective of this study is to evaluate the impact of clinical decision support (CDS) alert to notify providers when the opioid prescription being written will result in the patient transitioning into a new phase of opioid therapy. The 2022 CDC clinical practice guideline for prescribing opioids for pain recommends providers reassess patient pain as well as the risks and benefits of opioid therapy before patients transition from acute to subacute treatment (1 month of opioid analgesics) and when patients transition from subacute to chronic opioid treatment (3 months). This study will evaluate a clinical decision support tool identifying patients who will be transitioning between phases as a result of an opioid prescription and suggest a review of patient pain and goals. Primary care providers will be randomized at the clinic location to a control arm or intervention arm. The control arm will not be notified that the prescription transitions the patient to a new phase but will have access to the same patient pain scales and information. The intervention arm will receive a notification of the transition and suggest review of patient needs and encourage documentation. Opioid transition orders and outcomes of patients will be examined based on medical records data collected during routine care.

ELIGIBILITY:
Inclusion Criteria: Any primary care encounter where an opioid is prescribed that transitions the patient to a different stage of opioid therapy (acute to subacute after 1 month of opioids; subacute to chronic after 3 months of an opioid)

Exclusion Criteria:

* Patients <12 and >89
* Patients with active cancer diagnosis in last 1 year
* Patients with hospice care/palliative care order
* Patients with sickle cell disease diagnosis

Ages: 12 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents and visitors to the state of Colorado who seek healthcare within the University of Colorado Health (UCHealth) primary care system and receive an opioid prescription.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of encounters with an opioid transitioning prescription | 18 months
  The number of primary care encounters where an opioid prescription transitions a patient to a different phase of care (by phase) divided by the total number of opioid prescriptions

SECONDARY OUTCOMES:
Clinical decision support (CDS) acceptance rate | 18 months
  The number of times providers accepted the Clinical decision support (CDS) tool and documented a review of patient pain and goals
Subsequent opioid overdose/poisoning rates | Six months after an encounter where the opioid use disorder is identified
  The number of patients who reached the threshold of chronic opioid use, had a diagnosis of opioid overdose/poisoning or a new diagnosis of opioid use disorder
Opioid prescription abandonment | 18 months
  The proportion of opioid prescriptions initiated (triggering the CDS) and an opioid was not signed by the provider, indicating a change in clinical decision to prescribe an opioid
Number of patients with long term opioid use | Six months after an encounter where the opioid use disorder is identified
  Count of patients receiving >90 day supply of opioids

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hoppe, DO, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative EHR data utilized in this project will be housed on the National Addiction and HIV Data Archive Program (NAHDAP) website.
Supporting Information: Study Protocol
Time Frame: Data will be provided to NAHDAP after study results are published in peer-reviewed journals.
Access Criteria: Prior to downloading study data, the individual will have to register with the site and agree to a standard data use agreement.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/